CLINICAL TRIAL: NCT06237166
Title: Evaluation of an Online Intervention for Female Sexual Dysfunction: Randomized Controlled Trial
Brief Title: Evaluation of an Online Intervention for Female Sexual Dysfunction
Acronym: FELYCIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: Medical School Hamburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mylovia RCT
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Female Sexual Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mylovia + TAU (Experimental): Participants allocated to the intervention group will receive access to mylovia in addition to treatment as usual (TAU).
  mylovia is a digital health application designed for women with sexual dysfunction, accessible through a web browser. The application focuses on treatment methods derived from cognitive behavioral therapy (CBT). Topics addressed by mylovia are psychoeducation, relaxation and mindfulness exercises, strategies to improve self-esteem, development of passionate attitudes and situations, dealing with differences in desire in a relationship, and sensate focus exercises.
  The program operates through interactive "dialogues", which are accompanied by illustrations, audio recordings, motivational text messages, worksheets, and summaries. Users are also encouraged to regularly complete short questionnaires to monitor their complaints. Once registered, the program remains accessible for 180 days.
  Interventions: Behavioral: mylovia
- information material + TAU (No Intervention): Participants allocated to the control group will receive access to information material about treatment and counseling options in addition to treatment as usual (TAU).

INTERVENTIONS:
Behavioral: mylovia — Participants will receive access to the digital health intervention mylovia in addition to TAU.
  Arms: mylovia + TAU

SUMMARY:
In this randomized controlled clinical trial, 250 participants with female sexual dysfunction will be investigated regarding the effectiveness of an online intervention for improving sexual function, the unguided online intervention mylovia. Inclusion criteria are: female sex and female gender, age ≥18, diagnosed sexual dysfunction (ICD-11: HA00, HA01, HA02) or sexual pain disorder (ICD-11: HA20), low sexual functioning (<27 on the Female Sexual Function Index; FSFI), sufficient German skills, and consent to participation. Exclusion criteria are: biological, psychological or social factors that might interfere with study participation, and use of another digital intervention for sexual problems. Participants will be randomized and allocated to either an intervention group, receiving access to mylovia in addition to treatment as usual (TAU), or a control group, receiving information material about treatment and counseling options in addition to TAU. Primary endpoint will be sexual functioning assessed via FSFI, with three months post-allocation being the primary time point for assessment of effectiveness. Six months post allocation will be used as a timepoint for follow-up assessment of endpoints. Secondary endpoints will be sexual desire, sexual satisfaction, sexual pain, and general psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* female gender
* age ≥ 18 years
* diagnosis of sexual dysfunction (ICD-11: HA00, HA01, HA02) or sexual pain disorder (ICD-11: HA20), diagnosed via the DISEX-F interview
* Sexual function score (cut-off) of <27 on the FSFI
* consent to participation
* sufficient knowledge of the German language

Exclusion Criteria:

* Use of another digital intervention for sexual problems

In general, given that sexual dysfunction is a biopsychosocial phenomenon, mylovia is hypothesized to help women irrespective of the disorder's etiology (i.e., biological, psychological, or social). However, if one of the domains is extremely compromised, mylovia might not be expedient. Therefore, a clinical assessment of factors that might interfere with study assessment will be conducted, with the following additional exclusion criteria:

* Biological factors that might interfere with study participation (e.g., cancer, multiple sclerosis)
* Psychological factors that might interfere with study participation (e.g., schizophrenia, bipolar disorder, borderline personality disorder, eating disorder, post-traumatic stress disorder, severe depression, suicidality, substance use disorder)
* Social factors that might interfere with study participation (e.g. severe partnership problems)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — both female sex and female gender
Enrollment: 252 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
sexual functioning | 3 months
  Female Sexual Function Index (FSFI). Total score ranging from 2-36; higher scores mean better sexual function (better outcome).

SECONDARY OUTCOMES:
Depressive symptoms | 3 months, 6 months
  Patient Health Questionnaire - 9 item version (PHQ-9). Total score ranging from 0-27; higher scores mean more depressive symptomatology (worse outcome).
Sexual desire | 3 months, 6 months
  Sexual Interest and Desire Inventory - Female - Self-Report (SIDI-F-SR). Total score ranging from 0-51; higher scores mean higher levels of sexual desire (better outcome).
Sexual satisfaction | 3 months, 6 months
  New Sexual Satisfaction Scale - Short Form (NSS-SF). Total score ranging from 12 to 60; higher scores mean higher sexual satisfaction.
Sexual functioning | 6 months
  Female Sexual Function Index (FSFI). Total score ranging from 2-36; higher scores mean better sexual function (better outcome).

OTHER OUTCOMES:
Cognitions and behaviors related to sexual pain | 3 months, 6 months
  Self-compiled instrument assessing cognitions and behaviors related to sexual pain. Total score ranging from 0-100; higher scores mean more maladaptive cognitions and behaviors related to sexual pain (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Schröder, PhD, Principal Investigator — Medical School Hamburg
Locations (1):
- GAIA, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blaszcyk W, Buttner M, Betz LT, Riepenhausen A, Jacob GA, Klein JP, Schroder J. Digital intervention mylovia improves sexual functioning in women with sexual dysfunction in randomized controlled trial. NPJ Digit Med. 2026 Feb 3;9(1):115. doi: 10.1038/s41746-026-02385-z. PMID 41634129